CLINICAL TRIAL: NCT00221624
Title: Randomized Placebo-Controlled Trial of a Triple Therapy Combining Peginterferon Alfa-2a Plus Ribavirin Plus Amantadine Versus Peginterferon Alfa-2a Plus Ribavirin Plus Placebo in Hepatitis C-Infected Patients Non Responders to a First-Line Therapy of Interferon and Ribavirin
Brief Title: Peginterferon Alfa-2a Plus Ribavirin Plus Amantadine for the Treatment of Hepatitis C Infected Patients
Acronym: PEGARI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Hoffmann-La Roche (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7929-01; 2000-030
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2007-06-13 (Estimated); Status verified 2007-06

CONDITIONS: HCV Infection; Hepatitis C, Chronic
Keywords: Hepatitis C, chronic; HCV infection; Treatment failure; PEG Interferon; (Interferons/therapeutic use; Interferon Alfa-2a/adverse effects); ribavirin; (Ribavirin/therapeutic use; Ribavirin/adverse effects); Amantadine; Drug Therapy, Combination
MeSH Terms: conditions — Hepatitis C; Hepatitis C, Chronic | interventions — peginterferon alfa-2a; Ribavirin; Amantadine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Peginterferon alfa-2a
Drug: ribavirin
Drug: amantadine

SUMMARY:
Response to a second-line anti-HCV treatment in non responder patients to a first-line dual therapy remains very poor. Preliminary studies of amantadine suggest that this drug could be potentially effective to treat hepatitis C.

DETAILED DESCRIPTION:
Background : Response to a second-line anti-HCV treatment in non responder patients to a first-line dual therapy remains very poor. Preliminary studies of amantadine suggest that this drug could be potentially effective to treat hepatitis C.

Design : randomized, double-blind, multicenter trial.

Interventions compared : Peg-interferon alfa 2A + ribavirin + amantadine versus Peg-interferon alfa 2A + ribavirin + Placebo

Eligibility criteria : Chronic hepatitis C, previously treated with combination of interferon plus ribavirin for at least 24 weeks,detectable HCV RNA.

primary outcome : sustained virological response, defined as an undetectable HCV RNA level 24 weeks after the end of anti HCV treatment.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis C
* Previously treated with a combination of interferon plus ribavirin for at least 24 weeks
* Detectable HCV RNA (i.e. non responders)
* Signed informed consent

Exclusion Criteria:

* Evidence of another cause of liver disease
* Liver cirrhosis (child-Pugh stage BMC)
* Alcohol consumption > 30g/day for women or > 40g/day for men ; drug abuse
* Other serious relevant disorders : psychiatric condition (especially depression), cardio-vascular disease, renal decompensation, seizure history, hemoglobinopathy, auto-immune disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2001-11; Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
sustained virological response, defined as an undetectable HCV RNA level 24 weeks after the end of anti HCV treatment (i.e. overall 72 weeks after randomization) | 24 weeks after the end of antiHCV treatment

SECONDARY OUTCOMES:
ALT < upper limit of normal values, | 24 weeks after the end of anti-HCV treatment
histological response according to METAVIR score | 24 weeks after the end of anti-HCV treatment
adverse effects
quality of life assessed | at week 72

CONTACTS AND LOCATIONS:
Overall Officials: Patrice Couzigou, Pr, Principal Investigator — University Hospital, Bordeaux; Geneviève Chêne, Pr, Study Chair — University Hospital, Bordeaux
Locations (1):
- Service d'hépato-Gastro-Entérologie - Hôpital Haut Leveque - avenue de Magellan, Pessac, France